CLINICAL TRIAL: NCT01167387
Title: PREOPERATIVE ORAL CARBOHYDRATE LOADING: EFFECTS ON THE GLUCOSE METABOLISM AND POSTOPERATIVE INFECTIONS
Brief Title: Preoperative Carbohydrate Loading in Elective Surgery
Acronym: PROCY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: European Institute of Oncology (Other); San Raffaele University Hospital, Italy (Other); University of Siena (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Luca Vittorio Gianotti, professor of surgery, University of Milano Bicocca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROCY; SIS-E (Other Grant/Funding Number: SIS-E)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Surgery
Keywords: carbohydrate; glucose metabolism; surgery, outcome; major elective surgery; urology; hyperglicemia
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preoperative carbohydrate loading (Experimental): Patients in the treatment group will receive a carbohydrate beverage (total carbohydrates equal to 12.6g/100 mL: 2.1 g monosaccharide, 10.0 g maltodextrine; 240 mOsm/L) in dose of 800 mL. Patients will be free to drink the beverage from the evening before the operation and up to 2 hours before the induction of anesthesia
  Interventions: Dietary Supplement: PREOP
- water (Placebo Comparator): The control group will receive plain water with the same volume and timing of treatment.
  Interventions: Other: water

INTERVENTIONS:
Dietary Supplement: PREOP — a carbohydrate beverage (total carbohydrates equal to 12.6g/100 mL: 2.1 g monosaccharide, 10.0 g maltodextrine; 240 mOsm/L) in dose of 800 mL
  Arms: preoperative carbohydrate loading
Other: water — The control group will receive plain water with the same volume and timing of treatment.
  Arms: water

SUMMARY:
Postoperative infectious morbidity remain the most frequent, threatening and costly event after major surgery. Maintenance of postoperative euglycemia might be a key factor to prevent such complications and given the preliminary data on the positive effect of carbohydrate load on glucose metabolism it might also be valuable in improving outcome. If this treatment will be proved effective on relevant outcome measure such as rate of infections, it might be used routinely and extensively because preoperative carbohydrates administration is cheap, simple and applicable by everyone in any surgical ward.

The aim of the trial is to evaluate if the normalization of blood glucose by means of preoperative oral administration of maltodextrine, in patients candidate to elective major surgery, may be effective in improve surgical morbidity.

ELIGIBILITY:
Inclusion Criteria:

* patients candidate for elective major (expected duration > 2 hrs) abdominal, urologic, and gynecologic surgery

Exclusion Criteria:

* diagnosis of diabetes mellitus,
* baseline plasma glucose level > 125 mg/dl,
* pancreatic resection,
* ASA score > 3,
* malnutrition (loss of weight greater than 10%),
* emergency surgery,
* documented gastro-esophageal reflux,
* corticosteroid therapy,
* ongoing infection,
* pregnancy,
* age < 18 years,
* denied written informed consent

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
rate of postoperative complications | 30 days

SECONDARY OUTCOMES:
rate of patients needing insulin treatment | 4 days
rate of total complications | 30 day after surgery
rate of patients needing antibiotic therapy | 30 days after surgery
rate of reopaeration | 15 days
rate of patients needing intensive care treatment | 15 days
length of hospital stay | 15 days

OTHER OUTCOMES:
At least one postoperative measurement of blood glucose > 110 mL/dL e < 140 | 15 days
At least one postoperative measurement of blood glucose > 140 mL/dL e < 180 | 15 days
Severity of complications | 30 days
  grading according to Clavien
Duration of intensive care treatment | 15 days
Duration of overall complications | 30 days
Duration of antibiotic therapy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: luca gianotti, MD, PhD, Principal Investigator — Milano-Bicocca University
Locations (1):
- San gerardo hospital, Monza, Italy

IPD SHARING:
Plan to Share IPD: Yes